CLINICAL TRIAL: NCT00139555
Title: Effects of Amlodipine/Benazepril in Reducing Left Ventricular Hypertrophy in Patients With High Risk Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCIB002FUS16
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hypertension; Left Ventricular Hypertrophy
Keywords: Hypertension; Left ventricular hypertrophy
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — benazepril

INTERVENTIONS:
Drug: amlodipine/benazepril

SUMMARY:
Left ventricular hypertrophy (LVH) increases the risk of cardiovascular morbidity and mortality in patients with high blood pressure, compared to those without LVH. Reduction of left ventricular mass (LVM) with antihypertensive agents is associated with improved clinical outcome. This study will evaluate the effects of amlodipine/benazepril in reducing LVM in patients with high risk hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Males or female patients ≥ 55 years of age
* LVH as confirmed by echocardiogram
* Patients with high risk hypertension, currently treated or already taking antihypertensive medication

Exclusion Criteria:

* Renal artery stenosis
* Symptomatic heart failure or known ejection fraction < 40%
* Myocardial infarction or stroke within 6 months
* Presence of cranial aneurysm clips, coronary artery metal stents and pacemakers
* Pregnant or lactating females
* Cancer within the last 5 years

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2004-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in left ventricular mass index after 52 weeks

SECONDARY OUTCOMES:
Change from baseline in left ventricular mass after 52 weeks
Change from baseline in diastolic function after 52 weeks
Change from baseline in aorta function assessed blood pressure measurements after 52 weeks
Change from baseline in markers of fibrosis and increased heart size after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Reichek N, Devereux RB, Rocha RA, Hilkert R, Hall D, Purkayastha D, Pitt B. Magnetic resonance imaging left ventricular mass reduction with fixed-dose angiotensin-converting enzyme inhibitor-based regimens in patients with high-risk hypertension. Hypertension. 2009 Oct;54(4):731-7. doi: 10.1161/HYPERTENSIONAHA.109.130641. Epub 2009 Aug 17. PMID 19687350